CLINICAL TRIAL: NCT05327530
Title: A Phase II, Multicenter, Randomized, Open Label, Parallel-Arm, Umbrella Study of Avelumab (MSB0010718C) in Combination With Other AntiTumor Agents as a Maintenance Treatment in Participants With Locally Advanced or Metastatic Urothelial Carcinoma Whose Disease Did Not Progress With First Line Platinum-Containing Chemotherapy (JAVELIN Bladder Medley)
Brief Title: A Study of the Safety and Efficacy of Various Combinations of Avelumab as Therapy in Locally Advanced or Metastatic Urothelial Carcinoma (JAVELIN Bladder Medley)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany; Gilead Sciences; Nektar Therapeutics (Unknown)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS100070_0119; 2021-003669-36 (EudraCT Number); 2023-510139-12-00 (EU CTIS Number)
Record Dates: First submitted 2022-04-05; First posted 2022-04-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced or Metastatic Urothelial Carcinoma
Keywords: Avelumab; Avelumab in combination; Bladder cancer; M6223 (anti-TIGIT antibody); PD-L1; Sacituzumab govitecan (Trop-2 antibody drug conjugate); NKTR-255 (IL-15 agonist)
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — avelumab; sacituzumab govitecan; NKTR-255

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A: Avelumab (Experimental)
  Interventions: Drug: Avelumab
- Group B: Avelumab + Sacituzumab Govitecan (Experimental)
  Interventions: Drug: Avelumab; Drug: Sacituzumab Govitecan
- Group C: Avelumab + M6223 (Experimental)
  Interventions: Drug: Avelumab; Drug: M6223
- Group D: Avelumab + NKTR-255 (Experimental)
  Interventions: Drug: Avelumab; Drug: NKTR-255

INTERVENTIONS:
Drug: Avelumab — Participants will receive avelumab intravenous infusion at a dose of 800 milligrams (mg) once every 2 weeks (Q2W) until unacceptable toxicity, withdraw consent or initiation of a new treatment.
  Other Names: MSB0010718C
Drug: Sacituzumab Govitecan — Participants will receive sacituzumab govitecan intravenous infusion at dose of 10 milligrams per kilogram (mg/kg) of body weight once a week (Q1W) on Day 1 and 8 of 21-day treatment cycles, in combination with avelumab 800 mg Q2W, until unacceptable toxicity, withdraw consent or initiation of a new treatment.
  Other Names: IMMU-132; Trodelvy™; GS-0132
  Arms: Group B: Avelumab + Sacituzumab Govitecan
Drug: M6223 — Participants will receive M6223 (anti-T cell-immuno-receptor with Ig and ITM domains [anti-TIGIT]) intravenous infusion at dose of 1600 mg Q2W in combination with avelumab 800 mg Q2W, until unacceptable toxicity, withdraw consent or initiation of a new treatment.
  Arms: Group C: Avelumab + M6223
Drug: NKTR-255 — Participants will receive NKTR-255 intravenous infusion at a dose of 3 micrograms per kilogram body weight (mcg/kg) once every 4 weeks (Q4W) in combination with avelumab 800 mg Q2W, until unacceptable toxicity, withdraw consent or initiation of a new treatment.
  Arms: Group D: Avelumab + NKTR-255

SUMMARY:
The purpose of this study is to assess the safety and efficacy of avelumab in combination with other anti-tumor agents as a maintenance treatment in participants with bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed, unresectable locally advanced or metastatic urothelial carcinoma. Both transitional cell and mixed transitional/non- transitional cell histologies are allowed, but transitional cell carcinoma must be the predominant histology
* Participants has documented Stage IIIA/IIIB with N1-N3, or Stage IV disease (per American Joint Committee on Cancer/International Union for Cancer Control Tumor Node Metastasis system, 8th edition) at the start of first line chemotherapy.
* The last dose of first line chemotherapy must have been received no less than 4 weeks, and no more than 10 weeks, prior to randomization in the present study
* Estimated life expectancy of at least 3 months
* Participants without progressive disease as per RECIST v1.1 guidelines following completion of 4 to 6 cycles of 1L chemotherapy. Eligibility based on this criterion will be determined by Investigator review of pre chemotherapy and post chemotherapy radiological assessments (CT/MRI scans).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Adequate hematological, hepatic, and renal function as defined in the protocol
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with prior immunotherapy with Interleukin-2 (IL-2), IL-15, interferon alfa (IFN-α), or an anti programmed death receptor-1 (PD-1), anti programmed death-ligand 1 (PD-L1), anti PD-L2, anti CD137, or cytotoxic T cell lymphocyte-4 (CTLA-4) antibody (including ipilimumab), anti TROP2, anti-T-cell-immuno-receptor with Ig and ITM domains (anti-TIGIT) any other antibody or drug specifically targeting T cell costimulation or immune checkpoint pathways, agents targeting Nectin-4, or any of the investigational drugs used in combination with avelumab.
* Participants with active infection 48 hours before randomization requiring systemic therapy
* Participants with known prior or suspected hypersensitivity to study drugs or any component in their formulations
* Participants with prior adjuvant or neoadjuvant systemic therapy within 12 months of randomization
* Participants with vaccination within 4 weeks of the first dose of study treatment and while on trial is prohibited except for administration of inactivated vaccines (for example, inactivated influenza vaccines) administered >= 2 weeks prior first dose of study treatment. All severe acute respiratory syndrome coronavirus (SARS-CoV-2) vaccines approved or authorized by local Health Authorities are allowed
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) Assessed by Investigator | Time from randomization of study drug until first documentation of progressive disease (PD) or death, assessed approximately up to 51 months
Number of Participants with Treatment Emergent Adverse Events (TEAEs), Treatment-Related Adverse Events, and AEs of Special Interest (AESIs) as per Qualitative Toxicity Scale [National Cancer Institute-Common Terminology Criteria for Adverse Events 5.0] | From Randomization up to the last safety follow-up visit at approximately up to 51 months

SECONDARY OUTCOMES:
Overall Survival (OS) | Time from randomization of study drug until death, assessed approximately up to 51 months
Objective Response (OR) According to Response Evaluation Criteria in Solid Tumor (RECIST) v1.1 Assessed by Investigator | Time from randomization of study drug up to 51 months
Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumor (RECIST) v1.1 Assessed by Investigator | Time from first documented objective response to PD or death due to any cause, assessed approximately up to 51 months
Pharmacokinetic Serum Concentration of Avelumab, M6223, Sacituzumab govitecan and NKTR255 | Pre-dose up to safety follow up, assessed approximately up to maximum 51 months
Number of Participants with Positive Anti-Drug Antibody (ADA) of Avelumab, M6223, Sacituzumab govitecan and NKTR-255 | Baseline up to 51 months
Change From Baseline in National Comprehensive Cancer Network- Functional Assessment of Cancer Therapy (NCCN-FACT) Bladder Symptom Index- 18 (FBlSI-18) Disease Related Symptoms-Physical Subscale (DRS-P) Scores | Baseline, Week 13

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (97):
- United States (8):
  - Beacon Cancer Care, Coeur d'Alene, Idaho
  - University of Kansas Medical Center Research Institute, Inc. - 3901 Rainbow (MAIN), Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - AMR Kansas City, Formerly Center for Pharmaceutical Research, an AMR company - Kansas City, MO at St. Joseph Medical Center, Kansas City, Missouri
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Multicare Health System Tacoma General Hospital, Tacoma, Washington
  - University of Wisconsin Cancer Center, Madison, Wisconsin
- Australia (8):
  - Flinders Medical Centre, Bedford Park
  - Sunshine Hospital - PARENT, Footscray
  - Ashford Cancer Centre Research, Kurralta Park
  - Liverpool Hospital - PARENT, Liverpool
  - Calvary Mater Newcastle - PARENT, Newcastle
  - Tasman Oncology Research Ltd - Oncology, Southport
  - Macquarie University Hospital - PARENT, Sydney
  - The Kinghorn Can Cen, Westmead
- Belgium (8):
  - ZNA Middelheim - Middelheim - account 2, Antwerp
  - AZ Klina - PARENT, Brasschaat
  - Institut Jules Bordet - Medical Oncology, Brussels
  - Universitair Ziekenhuis Gent - Medical Oncology, Ghent
  - AZ Groeninge - Campus Kennedylaan - account 2, Kortrijk
  - Centre Hospitalier de l'Ardenne - PARENT, Libramont
  - CHU de Liège - PARENT, Liège
  - Universitaetsklinikum Wuerzburg - Klinik u. Poliklinik f. Urologie u. Kinderurologie, Wuerzburg
- Canada (4):
  - William Osler Health System - Brampton Civic Hospital, Brampton
  - CISSS de la Monteregie-Centre - Hospital Charles Le Moyne, Greenfield Park
  - CHUM Centre de Recherche, Montreal
  - The Ottawa Hospital Cancer Centre, Ottawa
- France (15):
  - Hôpital Foch - Service d'Oncologie Médicale, Suresnes, Hauts De Seine
  - ICO - Site Paul Papin - service d'oncologie medicale, Angers
  - Institut Bergonié - Service d'Oncologie Médicale, Bordeaux
  - Centre François Baclesse - Pathologies Gynecologiques, Caen
  - Hôpital Henri Mondor - Service d'Oncologie Médicale, Créteil
  - Clinique Victor Hugo - Centre Jean Bernard - Service d'Oncologie Médical, Le Mans
  - Centre Leon Berard - Service d'Oncologie Medicale, Lyon
  - Hôpital de la Timone - service d'urologie, Marseille
  - Hopital Caremeau - Service Hématologie Clinique/Oncologie Médicale, Nîmes
  - Hôpital Cochin - Hematologie et Oncologie Médicale, Paris
  - CHU Poitiers - Hôpital la Milétrie - service d'oncologie médicale, Poitiers
  - CRLCC Eugene Marquis - Service d'Oncologie médicale, Rennes
  - ICO - Site René Gauducheau - Service d'Oncologie medicale, Saint-Herblain
  - Clinique Sainte-Anne - Service d'Oncologie Médicale, Strasbourg
  - Institut de Cancérologie de Strasbourg Europe - ICANS - Service d'oncologie médicale, Strasbourg
- Germany (8):
  - Kliniken Maria Hilf GmbH - Klinik fuer Urologie, Muenchen, North Rhine-Westphalia
  - Universitaetsklinikum Halle (Saale) - Universitaetsklinik und Poliklinik fuer Urologie, Halle, Saxony-Anhalt
  - Universitaetsklinikum Essen - Westdeutsches Tumorzentrum, Essen
  - Universitaetsklinikum Frankfurt Goethe-Universitaet - Urologie und Kinderurologie2, Frankfurt
  - Universitaetsklinikum Wuerzburg - Klinik u. Poliklinik f. Urologie u. Kinderurologie, Halle
  - Kliniken Maria Hilf GmbH - Klinik fuer Urologie, Mönchengladbach
  - Universitaetsklinikum Muenster - Klinik und Poliklinik fuer Urologie, Münster
  - Universitaetsklinikum Tuebingen - Klinik fuer Urologie, Tübingen
- Greece (4):
  - Athens Medical Center, Athens
  - General Hospital of Athens "Alexandra", Athens
  - University General Hospital "Attikon", Athens
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
- Italy (14):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS - Oncologia Medica, Bologna
  - Azienda Ospedaliera Universitaria Careggi - S.O.D. di Oncologia Medica, Florence
  - IRCCS Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori "Dino Amadori" - IRST - Oncologia, Forlì
  - Fondazione IRCCS Istituto Nazionale dei Tumori - S.S. Oncologia Medica Genitourinaria, Milan
  - Ospedale San Raffaele - U.O. di Oncologia Medica, Milan
  - Humanitas Istituto Clinico Catanese - Oncologia Medica, Misterbianco
  - Istituto Nazionale Tumori Fondazione G. Pascale - Oncologia Medica A, Napoli
  - Istituto Nazionale Tumori Regina Elena IRCCS - Urologia, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS - U.O. Oncologia Medica 1, Padua
  - Azienda Ospedaliero Universitaria Pisana - U.O. Oncologia, Pisa
  - Ospedale Santa Maria delle Croci, Ravenna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Oncologia Medica, Rome
  - IRCCS Ospedale Casa Sollievo della Sofferenza - Dipartimento di Oncologia Medica, San Giovanni Rotondo
  - Azienda Ospedaliera S. Maria Di Terni - S.C. Oncologia Medica, Terni
- South Korea (8):
  - Chungnam National University Hospital - Department of Internal Medicine (Rheumatology), Daejeon
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (10):
  - Hospital Infanta Cristina - Unidad de Fase I, Badajoz
  - Hospital Clinic de Barcelona - Servicio de Oncologia, Barcelona
  - Hospital de la Santa Creu i Sant Pau - Dept of Oncology, Barcelona
  - Hospital del Mar - Servicio de Oncologia, Barcelona
  - Hospital Universitario Virgen del Rocio - Oncology Service, Barcelona
  - Hospital Universitario Reina Sofia - Dept of Oncology, Córdoba
  - Hospital General Universitario de Elche - Servicio de Oncologia, Elche
  - Hospital Universitario Lucus Augusti - Oncology, Lugo
  - Hospital General Universitario Gregorio Marañon - Servicio de Oncologia Medica, Madrid
  - ALTHAIA, Xarxa assistencial Universitaria de Manresa - Oncology Dept, Manresa
- Taiwan (7):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chi Mei Hospital, Liouying, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital,Linkou, Taoyuan District
- United Kingdom (3):
  - Barts Hospital - Dept of Medical Oncology, London, Greater London
  - The Christie Hospital - Dept of Oncology, Manchester
  - Royal Preston Hospital - Rosemere Cancer Centre, Preston

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Derived] Naing A, McKean M, Tolcher A, Victor A, Hu P, Gao W, Nogueira Filho MAF, Kitzing T, Gleicher S, Holland D, Richter E, Tadjalli-Mehr K, Siu LL. TIGIT inhibitor M6223 as monotherapy or in combination with bintrafusp alfa in patients with advanced solid tumors: a first-in-human, phase 1, dose-escalation trial. J Immunother Cancer. 2025 Feb 10;13(2):e010584. doi: 10.1136/jitc-2024-010584. PMID 39929671
- [Derived] Hoffman-Censits J, Grivas P, Powles T, Hawley J, Tyroller K, Seeberger S, Guenther S, Jacob N, Mehr KT, Hahn NM. The JAVELIN Bladder Medley trial: avelumab-based combinations as first-line maintenance in advanced urothelial carcinoma. Future Oncol. 2024 Feb;20(4):179-190. doi: 10.2217/fon-2023-0492. Epub 2023 Sep 6. PMID 37671748
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS100070_0119
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html